CLINICAL TRIAL: NCT01055873
Title: Immunology of the Infection Perinatal
Acronym: EP38
Status: Completed | Type: Observational
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Institut Pasteur (Industry); University of Paris 5 - Rene Descartes (Other); Hôpital Necker-Enfants Malades (Other)
Responsible Party: Lucie Marchand/Project manager, French National Agency for Research on AIDS and Viral Hepatitis
Other Study IDs: 2006-AO142-49
Record Dates: First submitted 2009-12-24; First posted 2010-01-26 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: HIV Infections
Keywords: immune status; adolescents or young adults infected; impact of viral replication
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: A single blood sample (30 mL) — A single blood sample (30 mL) was drawn during a hospital visit for clinical follow-up. Immunological assays were performed on fresh blood. Cells and plasma were stored and kept frozen for additional biological evaluations

SUMMARY:
ANRS-EP38-IMMIP is a non interventional study. A single blood sample (30 mL) was drawn during a hospital visit for clinical follow-up. Immunological assays were performed on fresh blood. Cells and plasma were stored and kept frozen for additional biological evaluations.

Patients are included in the French perinatal cohort (ANRS CO-10), or have been followed since before 1996 in the same clinical sites as patients who belong to ANRS CO-10. In the ANRS CO-10 cohort, all patients are prospectively followed from birth.

DETAILED DESCRIPTION:
Purpose:

Efficient anti-retroviral treatments lead to a significantly increased life expectancy. Children with perinatal infection are now reaching adulthood. The deleterious impact of viral replication during ontogenesis of the immune system, and the high thymic activity during the early years of life, preclude an extrapolation from data pertaining to the adult immune status and mean that specific pediatric studies are required. No data are available concerning the immune status of adolescents or young adults infected via materno-foetal transmission.

Detailed description:

Our assumption is that the duration of uncontrolled viral replication will affect the immune status after treatment because viral replication is associated with:

1. disease progression independently of CD4+ T cell levels;
2. accelerated senescence of the immune system;
3. destruction of organs involved in the restoration of major immune cell populations.

The aims of the study are:

1. to describe the immune and virological status of perinatally infected patients that are above 15 yrs old and
2. to study their associations with :

   1. the current virological/clinical and therapeutic status,
   2. the duration of uncontrolled viremia (defined by treatment history),
   3. the virological, immunological (CD4+ numbers), and clinical status at time of HAART initiation.

The immune status will be defined by (1) the number and phenotype of CD4+ and CD8+ T lymphocytes, dendritic cells, regulatory T cells, and NK cells, (2) the functions (proliferation and cytokine production) of CD4+ and CD8+ lymphocytes that are specific for HIV, a recall antigen (tetanus toxoid) and other viruses (CMV, EBV and Flu),the repertoire of Natural Killer cell receptors.

The virological status will be defined by the level of HIV DNA in PBMCs, the HIV subtype, resistance mutations in archived and circulating virus and sequences of the regions of the viral envelope involved in co-receptor use.

Clinical, therapeutic, demographic, virological and immunological data are collected from birth for members of the ANRS CO-10 cohort, and will be collected retrospectively since diagnosis for non-included patients.

ELIGIBILITY:
Inclusion criteria

* Being included in the ANRS CO-10 cohort, or being followed in the same sites as such patients since before 1996
* Being followed in the Paris area
* HIV-1 infected through the perinatal route, and not HIV-2 co-infected
* No therapeutic changes for at least 6 months; single molecule change without modification of viral load is tolerated.
* Informed consent signed by the patients and by their legal guardians for those younger than 18.
* Being affiliated to the Exclusion criteria French national social security system

Exclusion criteria

- Not Being affiliated to the French national social security system

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are included in the French perinatal cohort (ANRS CO-10), or have been followed since before 1996 in the same clinical sites as patients who belong to ANRS CO-10. In the ANRS CO-10 cohort, all patients are prospectively followed from birth
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2007-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To describe the immune and virological status of perinatally infected patients that are above 15 yrs old and

SECONDARY OUTCOMES:
To study their associations with the current virological/clinical and therapeutic status, the duration of uncontrolled viremia (defined by treatment history), the virological, immunological (CD4+ numbers), and clinical status

CONTACTS AND LOCATIONS:
Overall Officials: Warszawski MD Josiane, Methodologist, Study Chair — INSERM U 822, Hôpital de Bicêtre, portes 10 à 15, 82 rue du Général Leclerc, 94276 Le Kremlin-Bicêtre Cedex warszaws@vjf.inserm.fr ; Tel : 01 45 21 22 86; Blanche PHD Stéphane, Principal Investigator — Hopital Necker Enfants malades-Service immunologie hématologie pédiatrique -149 rue de Sèvres- 75015 PARIS 01 44 49 48 24

REFERENCES:
- [Derived] Avettand-Fenoel V, Blanche S, Le Chenadec J, Scott-Algara D, Dollfus C, Viard JP, Bouallag N, Benmebarek Y, Riviere Y, Warszawski J, Rouzioux C, Buseyne F. Relationships between HIV disease history and blood HIV-1 DNA load in perinatally infected adolescents and young adults: the ANRS-EP38-IMMIP study. J Infect Dis. 2012 May 15;205(10):1520-8. doi: 10.1093/infdis/jis233. Epub 2012 Mar 15. PMID 22427678
- See also: Related Info — http://www.anrs.fr